CLINICAL TRIAL: NCT05884853
Title: The Plasticity of Social Brain Network in Adults With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202012163RIND
Record Dates: First submitted 2023-05-04; First posted 2023-06-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: 40 autistic adolescents are recruited with their care givers. Also, 40 healthy controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD group (Experimental): autistic adolescents with their caregiver
  Interventions: Behavioral: PEERS
- Control group (Sham Comparator): healthy control without their caregiver
  Interventions: Behavioral: PEERS

INTERVENTIONS:
Behavioral: PEERS — The Program for the Education and Enrichment of Relational Skills (PEERS®) studies is an evidence-based 16-week group-based social skill training program developed for adolescents and young adults with ASD.

SUMMARY:
"Social brain" refers to brain regions dedicated to processing social information and enabling us to recognize and evaluate others' mental states. The social brain hypothesis suggests that our brains evolve to navigate complex social systems. The social brain is hypothesized to consist of a distributed network including the posterior superior temporal sulcus (pSTS), the dorsal and ventral medial prefrontal cortices (dmPFC and vmPFC), ACC and posterior cingulate cortex (PCC), the amygdala, the orbital frontal cortex (OFC), and the fusiform gyrus (FG), TPJ, inferior occipital gyrus (IOG), and the insula. Each region serves distinct role while works together to support social processing, including perceiving, interpreting, and generating responses to the intentions, dispositions, and behaviors of others.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50
* diagnosed with ASD from licensed mental health or medical professional based on DSM5
* have social problems
* motivated to participate in the treatment
* fluent in chinese
* caregiver also fluent in chinese and motivated to participate
* had a full-scale IQ > 70 on WAIS-IV
* scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ), indicating clinical impairment associated with ASD.

Exclusion Criteria:

* history of major mental illness, such as bipolar affective disorder, schizophrenia, psychosis, or neurological diseases
* visual impairment and/or hearing impairment
* any metal, electronic part that cannot be removed from the body, or being pregnant, which may not be able to use fMRI scan.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Interview Revised, ADIR | 16 weeks
  Interview of the caregivers that covers most developmental and behavioral aspects of ASD. Range from 0 to 8, higher the score, worse the symptom.
The Autism Diagnostic Observation Schedule, ADOS | 16 weeks
  Diagnosing and assess autism. Range from 0 to 8, higher the score, worse the symptom.
Autism Spectrum Quotient | 16 weeks
  50 items, total score range from 0 to 50. Higher the score, worse the symptom
Social Responsiveness Scale, Second Edition (SRS-2) | 16 weeks
  65 items, total score range from 65 to 260. Higher the score, worse the symptom
Quality of Socialization Questionnaire (QSQ) | 16 weeks
  12 items, total score range from 0 to 12.Higher the score, better the frequency and quality of socialization
The Empathy Quotient (EQ) | 16 weeks
  40 items, total score range from 0 to 80. Higher the score, worse the empathy

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan